CLINICAL TRIAL: NCT02309489
Title: Involving Men in Maternity Care in Burkina Faso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Strengthening Evidence for Programming on Unintended Pregnancy (STEP UP) (Unknown); Department for International Development, United Kingdom (Other Government); Economic and Social Research Council, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QA649
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2016-09

CONDITIONS: Postpartum Period
Keywords: Family Planning Services; Maternal Health Services; Breast Feeding; Contraception; Postnatal care; Postpartum contraception; Exclusive breastfeeding; Postpartum Period
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): * Receive standard maternity care
  * Woman and partner attend one extra couple counselling session during pregnancy (A)
  * Partner attends one group education session for men (B)
  * Partner participates in pre-discharge consultation (C)
  Interventions: Behavioral: Partner involvement
- Control (No Intervention): * Receive standard maternity care
  * No active encouragement of partner involvement, no extra sessions offered

INTERVENTIONS:
Behavioral: Partner involvement — Partner is involved in maternity care
  Arms: Intervention

SUMMARY:
The uptake of postpartum contraception, postpartum care attendance and the practice of exclusive breastfeeding are low in Sub-Saharan Africa. Although the involvement of men in maternity care has been shown to be a promising strategy for the achievement of other reproductive health goals, little is known about the effect of their participation on these outcomes. This study aims to test whether the involvement of men can improve care-seeking and promote healthy behaviours among postpartum women in Burkina Faso.

DETAILED DESCRIPTION:
There is a paucity of evidence on strategies to increase the uptake of postpartum contraception and attendance at facility-based postpartum care in developing countries, including in Sub-Saharan Africa. There is also a need to test new solutions to improve adherence to recommended infant feeding practices in these settings. Partner opposition is a major barrier to women's uptake of contraceptive methods in the postpartum period in Burkina Faso, and research has shown the need to sensitise and inform men about a broad range of topics related to reproductive health. However, the effect of involving male partners on women's and newborns' health and wellbeing in low-resource settings is not well known, and there is particularly little evidence for outcomes related to the postpartum period.

The aim of this study is to assess whether male partner involvement in maternity care has the potential to increase care-seeking and promote healthy behaviours among postpartum women in an urban West-African setting. A randomized controlled trial (RCT) of an intervention to promote the involvement in maternity care of the partners of pregnant women attending primary health care facilities will be conducted in the city of Bobo-Dioulasso. The intervention consists of three extra components in addition to standard maternity care: one extra couple counselling session during pregnancy (A), partner participation in a group education session for men (B), and partner participation in the pre-discharge consultation after birth (C). Women in the control group will receive standard maternity care only, in which men do not participate.

A qualitative component will be carried out alongside the RCT, in order to examine the factors that may have determined the success, or lack thereof, of the intervention by reflecting on the experience of participants (women, partners , and health workers), and to explore their attitudes, beliefs and concerns relative to partner involvement in maternity care, through focus group discussions and in-depth interviews.

The policy implications of the study findings will be assessed and, if appropriate, a strategy will be developed for their dissemination among policymakers and other stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-18, married, or
* Age 18+, in a co-habiting relationship
* Pregnant 24-36 weeks
* No obstetric risk factors requiring hospital delivery
* Lives no more than one hour away on foot, not planning to move from the city
* Gives informed consent

Exclusion Criteria:

* Not meeting inclusion criteria
* Declines to participate

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1144 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Daniele, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- District Sanitaire de Dafra, Bobo-Dioulasso, Burkina Faso

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: * Receive standard maternity care
  * Woman and partner attend one extra couple counselling session during pregnancy (A)
  * Partner attends one group education session for men (B)
  * Partner participates in pre-discharge consultation (C)
  Partner involvement: Partner is involved in maternity care
Period: Overall Study
Arm/Group | Intervention | Control
Started | 583 | 561
Follow-up at 3 Months Postpartum | 560 | 541
Completed (Follow-up at 8 months postpartum) | 568 | 547
Not Completed | 15 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 583 | 561 | 1144
Age, Customized [Count of Participants; unit: Participants]
  15-19 | 73 | 76 | 149
  20-24 | 179 | 164 | 343
  25-29 | 163 | 158 | 321
  30-34 | 109 | 99 | 208
  35-39 | 46 | 56 | 102
  40-45 | 13 | 9 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 583 | 561 | 1144
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Bobo, Bwa | 109 | 110 | 219
  Dagara, Lobi, Birifor, Djan, & similar | 61 | 41 | 102
  Dioula, Dafing, Samo, & similar | 93 | 85 | 178
  Gourounsi, Ko, Nounouma | 24 | 24 | 48
  Mossi, Gourmanche, Bissa, & similar | 260 | 263 | 523
  Peulh | 16 | 19 | 35
  Other | 21 | 15 | 36
Health centre of recruitment [Count of Participants; unit: Participants]
  Bolomakote | 89 | 86 | 175
  Guimbi | 101 | 109 | 210
  Ouezzinville | 163 | 165 | 328
  Sarfalao | 119 | 92 | 211
  Secteur 24 | 111 | 109 | 220
Religion [Count of Participants; unit: Participants]
  Muslim | 420 | 407 | 827
  Christian | 158 | 144 | 302
  Traditional/animist | 1 | 5 | 6
  No religion | 1 | 0 | 1
Education [Count of Participants; unit: Participants]
  No education | 311 | 278 | 589
  At most primary completed | 145 | 168 | 313
  Above primary | 126 | 115 | 241
Parity [Count of Participants; unit: Participants]
  No children | 127 | 144 | 271
  1 child | 159 | 132 | 291
  2 children | 119 | 93 | 212
  3 children or more | 178 | 192 | 370

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Attending the Recommended Number of Postnatal Care Appointments
Description: This was defined as whether women had attended at least two outpatient postnatal care consultations/check-ups in the first six weeks after birth.
Time Frame: Data collected at 3 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 560 | 541
Participants | 342 | 265

2. Primary Outcome: Number of Participants Practicing Exclusive Breastfeeding at 3 Months Postpartum
Description: This was defined according to the WHO criteria for exclusive breastfeeding: "the infant has received only breastmilk from his/her mother or a wet nurse, or expressed breastmilk, and no other liquids or solids with the exception of drops or syrups consisting of vitamins, mineral supplements or medicines". Although the WHO recommends exclusive breastfeeding for the first 6 months postpartum, 3 months was chosen as the reference period because by that point only 20% of infants are still exclusively breastfed.
Time Frame: Data collected at 3 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 535 | 511
Participants | 232 | 161

3. Primary Outcome: Number of Participants Using Effective Modern Contraception at 8 Months Postpartum
Description: Effective modern methods were defined as those having a rate of unintended pregnancy per 100 women of 10% or less per year, as commonly used. Based on local availability, these methods were: implants, IUDs, injectables, oral contraceptives, and permanent methods. Each woman was considered a "user" or "non-user" for each method.
Time Frame: Data collected at 8 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 554 | 533
Participants | 330 | 283

4. Secondary Outcome: Number of Participants Using Long Acting or Permanent (LA/PM) Methods of Contraception at 8 Months Postpartum
Description: This was defined as the number of women using IUDs, implants, female sterilization or male sterilization at 8 months postpartum.
Time Frame: Data collected at 8 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 554 | 533
Participants | 170 | 122

5. Secondary Outcome: Number of Participants Using Any Contraceptive Method at 8 Months Postpartum
Description: This was defined as the use of all contraceptive methods, according to self-report at 8 months postpartum. The aim of this measure was to quantify the use of "natural" methods, such as withdrawal, which, based on the literature, may be higher than reported in DHS surveys.
Time Frame: Data collected at 8 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 554 | 533
Participants | 391 | 343

6. Secondary Outcome: Number of Participants Who Initiated Postpartum Contraception in a Timely Fashion
Description: Whether or not users of modern contraception at 8 months postpartum had initiated their method in a timely fashion was assessed. This was a binary outcome with users of effective methods as the denominator. Users were considered to have initiated contraception either in a timely fashion, or not in a timely fashion. Timeliness in this context refers to whether women had been exposed to a significant risk of becoming pregnant prior to initiating their contraceptive method.
  Specifically, whether or not women using contraception had initiated it in a timely fashion ("timeliness") was defined based on the interaction between four criteria: when they initiated the method (either in the first 6 months postpartum or later); whether they had reported to be exclusively breastfeeding at 3 months postpartum (yes or no); whether at that point in time they had resumed intercourse (yes or no); and whether at that point their menses had returned (yes or no).
Time Frame: Data collected at 8 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 329 | 281
Participants | 249 | 188

7. Secondary Outcome: Number of Participants With an Unmet Need for Contraception at 8 Months Postpartum
Description: Unmet need for contraception is a concept used to describe the situation in which women are at risk of conceiving, yet do not wish to become pregnant. Several definitions of unmet need for contraception have been proposed. The Revised definition of unmet need published by the DHS Program in 2012 was chosen. This definition classifies women as either having an unmet need, or not, based on the interaction of several criteria: whether or not they wanted the index pregnancy; whether or not their periods have returned after giving birth; whether or not they want to become pregnant again, and if so how soon.
Time Frame: Data collected at 8 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 560 | 539
Participants | 79 | 101

8. Secondary Outcome: Number of Participants With High Relationship Adjustment at 8 Months Postpartum
Description: Relationship adjustment, as defined in this study, was a score calculated based on questions related to: woman's self-reported satisfaction with the relationship; her level of communication and agreement with her male partner on issues related to reproductive health; and who in the household made decisions related to reproductive health and any relevant expenditures. The questions used were derived from similar survey measures (Spanier's Dyadic Adjustment Scale and the Locke-Wallace Marital Adjustment Test (LWMAT)). The median score was chosen as a cut-off point, above which women were considered to have high relationship adjustment, and below which they were considered to have low relationship adjustment.
Time Frame: Data collected at 8 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 568 | 457
Participants | 323 | 263

9. Other Pre Specified Outcome: Number of Participants With Complete Satisfaction With Care
Description: A tailored satisfaction score was developed to assess participant's satisfaction with routine maternity care received. Questions were adapted from the K4 Health's Respectful Maternity Care toolkit, and from the UK's Care Quality Commission (CQC)'s 2013 Maternity Services Survey. If participants reported having experienced the maximum score for each dimension of satisfaction, they were classed as having complete satisfaction with care.
Time Frame: Data collected at 3 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 560 | 541
Participants | 413 | 395

10. Other Pre Specified Outcome: Number of Participants in the Intervention Group With High Adherence to the Intervention
Description: High adherence to the intervention was defined as attendance (by the couple or the partner) at at least two out of three intervention components.
Time Frame: Process data collected throughout intervention implementation
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 583
Participants | 432

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed during each phase of data collection (baseline interviews, 3-month postpartum follow-up interviews, and 8-month postpartum follow-up interviews).
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 2/583 | 1/561
Serious Adverse Events (participants affected / at risk) | 0/583 | 0/561
Other Adverse Events (participants affected / at risk) | 0/583 | 0/561

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No